CLINICAL TRIAL: NCT05488769
Title: Visual Outcomes and Patient Satisfaction After Bilateral Implantation of Non-diffractive EDOF IOL Made of a New Hydrophobic Acrylic Material
Status: Terminated | Type: Observational
Why Stopped: Investigational product not available
Sponsor: Thomas Nagy (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor-Investigator, Thomas Nagy, Principal Investigator, Vision North Eye Centre
Organization: Vision North Eye Centre (Other)
Other Study IDs: TN-22-001
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Clareon Vivity extended depth of focus (EDOF) intraocular lens: Implantation with the Clareon Vivity extended depth of focus (EDOF) intraocular lens
  Interventions: Device: Clareon Vivity extended depth of focus (EDOF) intraocular lens

INTERVENTIONS:
Device: Clareon Vivity extended depth of focus (EDOF) intraocular lens — Implantation with the Clareon Vivity extended depth of focus (EDOF) intraocular lens

SUMMARY:
The objective is to measure the range of vision and patient reported visual disturbances after bilateral implantation for this unique non-diffractive extended depth of focus (EDOF) intraocular lens (IOL) made from the Clareon material.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of binocular distance-corrected distance (6m) and intermediate (66cm) visual acuity after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include administration of a visual disturbance questionnaire (QUVID), and a satisfaction questionnaire (IOLSAT), as well as measurement of bilateral visual acuity and manifest refraction.

ELIGIBILITY:
Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Visually significant age-related cataracts bilaterally.
* Best monocular Corrected distance Visual Acuity predicted to be (20/25) or better after cataract removal and IOL implantation as determined by surgeon.
* Gender: Males and Females.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Clear intraocular media other than cataract.
* Planned Bilateral implantation of the Clareon Vivity and Vivity toric IOLs.
* IOL powers between 6D and 30D, T2-T6.

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Previous ocular or refractive surgery
* Ocular surface disease/Dry Eye Disease
* Intraoperative complications during procedure
* Glaucoma, including well-controlled
* Any disorders that reduce binocular vision (ie Strabismus)
* Any ocular comorbidity that, in the opinion of the investigator reduce post-op visual acuity (e.g. AMD etc)

The principal investigator reserves the right to declare a patient ineligible or non- evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Eligible test subjects will be presenting for cataract surgery who are interested in a reduced dependence on spectacles for intermediate and distance vision, and who are considered appropriate candidates for EDOF lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Binocular distance-corrected visual acuity at distance (6m) | 3 months postoperative
Binocular distance-corrected visual acuity at intermediate (66cm) | 3 months postoperative

SECONDARY OUTCOMES:
Percentage of eyes with absolute prediction error less than or equal to 0.50D | 3 months postoperative
Percentage of eyes with refractive astigmatism less than or equal to 0.50 D | 3 months postoperative

OTHER OUTCOMES:
Satisfaction questionnaire | 3 months postoperative
  The Intraocular Lens Satisfaction questionnaire (IOLSAT). Lower scores indicate higher spectacle independence and satisfaction.
Visual disturbances questionnaire | 3 months postoperative
  Questionnaire for Visual Disturbances (QUVID). Lower scores indicate less frequent, severe, or bothersome visual disturbances.
Binocular uncorrected and distance-corrected visual acuity at near (40cm) | 3 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nagy, MD, Principal Investigator — Vision North Eye Centre
Locations (1):
- Vision North Eye Centre, Terrace, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No